CLINICAL TRIAL: NCT03258372
Title: A Phase 1, Open-Label, Fixed-Sequence, Crossover Drug-Drug Interaction Study in Healthy Subjects to Determine the Effects of a Strong Inducer of Cytochrome P450 3A on Exposure to Mifepristone and Its Metabolites
Brief Title: Crossover Drug-Drug Interaction Study to Determine Effects of Cytochrome P450 3A on Exposure to Mifepristone and Its Metabolites
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Corcept Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: C1073-37
Record Dates: First submitted 2017-08-21; First posted 2017-08-23 (Actual); Last update posted 2018-02-23 (Actual); Status verified 2017-11

CONDITIONS: Healthy
MeSH Terms: interventions — Mifepristone; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): Mifepristone 300 MG, 1 tablet
  Interventions: Drug: Mifepristone
- Cohort 2 (Experimental): Mifepristone 1500 MG, 5 tablets
  Interventions: Drug: Mifepristone

INTERVENTIONS:
Drug: Mifepristone — Period 1: mifepristone 300 MG (1 tablet) for a total of 300 MG on Day 1 in Cohort 1; and mifepristone 300 MG (5 tablets) for a total of 1500 MG in Cohort 2; then Period 2: rifampin 300 MG (2 capsules) for a total of 600 MG daily for 14 days for both cohorts; then Period 3: mifepristone 300 MG (1 tablet) for a total of 300 MG on Day 1 in Cohort 1; and mifepristone 300 MG (5 tablets) for a total of 1500 MG in Cohort 2
  Other Names: rifampin

SUMMARY:
This is a Phase 1, single center, fixed sequence, open label, drug-drug interaction study of the effect of multiple doses of rifampin 600 mg daily, a strong CYP3A inducer, on the exposure of mifepristone at 2 dose levels.

ELIGIBILITY:
Inclusion Criteria:

* Be healthy
* Have a BMI of 18 to 32 kg/m2, inclusive, and body weight more than 50 kg (110 pounds)
* Be judged to be in good health, based on the results of medical history, physical examination, vital signs, 12-lead ECG, and clinical laboratory findings
* Have suitable veins for multiple venipuncture/cannulation
* Female subjects of childbearing potential must use highly effective contraception with low user-dependency. The only acceptable method is an intrauterine device (IUD), provided that the subject has tolerated its use for at least 3 months before the first dose of study drug and undertakes not to have it removed for 1 month after the last dose of study drug. Use of hormonal contraception (by any route, including intrauterine hormone releasing systems) or hormone replacement therapy is NOT acceptable.

Exclusion Criteria:

* Have multiple drug allergies, or be allergic to any of the components of mifepristone or rifampin
* Have a condition that could be aggravated by glucocorticoid blockade (eg, asthma, any chronic inflammatory condition)
* Have a history of unexplained vaginal bleeding, endometrial hyperplasia with atypia or endometrial carcinoma
* Breastfeeding
* In the 1 year before first study drug administration, have a history of drug or alcohol abuse
* In the 6 calendar months before first study drug administration, on average

  * Have smoked more than 5 cigarettes/day
  * Have consumed more than 21 units of alcohol/week for male subjects or 14 units for female subjects (1 unit/drink = 5 ounces of wine, or 12 ounces of beer, or 1.5 ounces of hard liquor)
* In the 2 calendar months before first study drug administration, have donated/lost blood or plasma in excess of 400 mL
* In the 30 days before first study drug administration, have participated in another clinical trial of a new chemical entity or a prescription medicine

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2017-08-16 (Actual); Primary Completion 2017-11-29 (Actual); Study Completion 2017-11-29 (Actual)

PRIMARY OUTCOMES:
Cmax of mifepristone of period 1 vs Cmax of mifepristone of period 3 | 18 days
  Maximum (peak) plasma drug concentration (Cmax)
AUC0-tz of mifepristone of period 1 vs AUC0-tz of mifepristone of period 3 | 18 days
  Area under the concentration-time curve from zero up to the last concentration above the lower limit of quantification of the assay (AUC0-tz)
AUCinf of mifepristone of period 1 vs AUCinf of mifepristone of period 3 | 18 days
  Area under the plasma concentration-time curve from time zero to infinity (AUCinf)

SECONDARY OUTCOMES:
Cmax of mifepristone metabolites of period 1 vs Cmax of mifepristone metabolites of period 3 | 18 days
AUC0-tz of mifepristone metabolites of period 1 vs AUC0-tz of mifepristone metabolites of period 3 | 18 days
AUCinf of mifepristone metabolites of period 1 vs AUCinf of minfepristone metabolites of period 3 | 18 days

CONTACTS AND LOCATIONS:
Overall Officials: Ada Lee, MD, Study Director — Corcept Therapeutics
Locations (1):
- SeaView Reserch, Miami, Florida, United States